CLINICAL TRIAL: NCT03304990
Title: Panomics Relationships in the Epidemiology of Cancer Through In Silico Expression (PRECISE)
Status: Withdrawn | Type: Observational
Why Stopped: PI has left our Inst.
Sponsor: Greater Baltimore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PRECISE
Record Dates: First submitted 2017-09-26; First posted 2017-10-09 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cancer; Patients With Clinical and Environmental Risk Factors for Cancer; Patients With a Suspected or Confirmed Diagnosis of Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Collection of saliva and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family History of CA: Hereditary cancer genetic screening based on risk factors
  Interventions: Other: Patients with CA or suspected risk of CA or a family Hx
- Risk Factors for CA: No dx of CA
  Interventions: Other: Patients with CA or suspected risk of CA or a family Hx
- Suspected or Confirmed Diagnosis of CA: Suspected or confirmed diagnosis of cancer
  Interventions: Other: Patients with CA or suspected risk of CA or a family Hx

INTERVENTIONS:
Other: Patients with CA or suspected risk of CA or a family Hx — Patients with Family History of Cancer, (ii) Patients with Clinical and Environmental Risk Factors for Cancer, (iii) Patients with a Suspected or Confirmed Diagnosis of Cancer.

SUMMARY:
PRECISE is a study to discover new detection, prognosis and treatment biomarkers for cancer. This is a prospective, multi-center, observational study designed to collect de-identified biospecimens and clinical data from a large cohort of participants from clinical research networks in the United States. In this study, the investigators propose creating a large-scale normalized panomics dataset specifically designed for deep learning-based in silico analysis for biomarker discovery.

DETAILED DESCRIPTION:
This study will enroll all subjects who are eligible and willing to participate with a goal of enrolling at least 10,000 in several categories: (i) Patients with Family History of Cancer, (ii) Patients with Clinical and Environmental Risk Factors for Cancer, and (iii) Patients with a Suspected or Confirmed Diagnosis of Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Family History of Cancer

  1. Ages 18 or older
  2. Either of the following:

     1. Patients with two or more first, second or third degree blood relatives on the same side of the family diagnosed with cancer
     2. Patients with one or more first, second or third degree blood relative with male breast cancer
     3. Patients with a first, second, or third degree blood relative with a known BRCA1 or BRCA2 mutation
     4. Patients with a first, second, or third degree blood relative who has had colorectal or endometrial cancer diagnosed before age 50 years
     5. Patients with first degree relatives with a known deleterious APC, MEN1, MUTYH, PTEN, RET, STK11, TP53, or VHL gene mutation
     6. Patients of Ashkenazi Jewish descent with one or more first degree relatives or two or more second degree relatives with breast, ovarian or colorectal cancer
  3. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form

     Patients with Clinical & Environmental Risk Factors for Cancer

  <!-- -->

  1. Either of the following:

     1. Women 21 or older
     2. Men 50-75
     3. Men 75-85, with a history of smoking
  2. At least one guideline recommended cancer screening test documented in the medical record, if indicated for age and gender (eg, pap smear, mammography, low dose chest CT and/or colonoscopy)
  3. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form Cancer Patients

  <!-- -->

  1. Ages 18 or older
  2. Either of the following:

     1. New diagnosis of histologically confirmed cancer (any stage I-IV, as well as carcinoma in situ (CIS)), across multiple solid tumor types with no prior systemic cancer therapy and scheduled for surgical resection or non-surgical management
     2. Or, subjects with a high suspicion for cancer diagnosis by clinical and radiological assessment, but without preceding histologic diagnosis, are eligible, if they have not received prior systemic cancer therapy and are scheduled for surgery
  3. Has or will have a medically obtained pathological tumor specimen from core needle or surgical biopsy and/or surgical resection within 4 weeks (28 days) of study blood draw and pre-treatment
  4. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form

Exclusion Criteria:

* 1. Blood or blood product transfusion in the preceding 2 months 2. Cognitive impairment as determined by clinical history 3. Pregnant women (by self-report of pregnancy status) 4. Inability to speak English 5. Previous diagnosis of cancer except: non-melanomatous skin cancer 6. Poor health status or unfit to tolerate blood draw

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with Family History of Cancer, whose immediate or extended family member(s) were diagnosed with cancer (20% of the Study Enrollment),
  * Patients with Clinical and Environmental Risk Factors for Cancer (20% of the Study Enrollment),
  * Patients with a Suspected or Confirmed Diagnosis of Cancer (60% of the Study Enrollment).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Panomics Relationships in the Epidemiology of Cancer through In Silico Expression (PRECISE) | 5 years
  * Establish and maintain a unique repository of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected from thousands of patients 18 years of age or older who have cancer or are at risk of developing cancer.
  * Discover and validate new detection, prognosis and treatment biomarkers for cancer
Panomics Relationships in the Epidemiology of Cancer through In Silico Expression (PRECISE) | 5 years
  ● Determine candidate genes and markers underlying cancer and response to treatment.
Panomics Relationships in the Epidemiology of Cancer through In Silico Expression (PRECISE) | 5 years
  ● Discover and validate new detection, prognosis and treatment biomarkers for cancer

CONTACTS AND LOCATIONS:
Overall Officials: Neri Cohen, Principal Investigator — Greater Baltimore Medical Center IRB
Locations (1):
- Greater Baltimore Medical Center, Baltimore, Maryland, United States